CLINICAL TRIAL: NCT01968538
Title: A Pilot Study to Establish a Standardized Protocol for Omic Analysis of Patients With Clinically Localized Prostate Cancer Receiving Radiation Therapy
Brief Title: Metabolomic Study for Localized Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-096
Record Dates: First submitted 2013-09-19; First posted 2013-10-24 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiosurgery; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimen:For future Research Optional Destruction if requested identifiable Urine yes no yes no Sputum yes no yes no Blood yes no yes no
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prostate Cancer Patients: Prostate cancer patients who underwent radiation therapy
  Interventions: Radiation: Radiation Therapy
- Healthy control: age-matched male who has no known prostate cancer

INTERVENTIONS:
Radiation: Radiation Therapy
  Other Names: Prostate stereotactic body radiation therapy (SBRT) and intensive modulated radiation therapy (IMRT) or the combination of both (boost)
  Groups: Prostate Cancer Patients

SUMMARY:
Prostate cancer is a common disease in men treated using surgery, radiation therapy and/or hormonal therapy. Clinical prognosis relates to stage and grade of disease. Recent advances in omic analysis may offer additional information to the physician about prognosis and radiation response. We propose to establish a protocol to incorporate omic analysis into the evaluation and treatment of patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males who are older than 18 years old,
* with clinically localized prostate cancer
* are receiving radiation therapy

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 prostate cancer patients vs. 200 healthy men
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-01; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
molecular changes in biofluid | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Collins, MD, PhD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Arlington, Virginia, United States